CLINICAL TRIAL: NCT04700644
Title: Assessment of Central Adrenal Insufficiency in Adults With Prader-Willi Syndrome.
Brief Title: Assessment of CAI in Adults With PWS.
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Magda Goralska, Principal Investigator, Medical University of Warsaw
Other Study IDs: CAIPWS
Record Dates: First submitted 2020-06-21; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Central Adrenal Insufficiency; Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: The prevalence and clinical significance of central adrenal insufficiency (CAI) in adult patients with Prader Willi Syndrome (PWS) remains unclear.

Aim: To assess the prevalence of CAI in adults with PWS and to analyse the effects of replacement therapy with hydrocortisone (HCT) in patients with suspected CAI.

Material and Methods: Twenty one adult patients with PWS were evaluated. Based on peak cortisol at the 30 minute of the high dose short Synacthen test (HDSST), patients were divided into three groups: CAI (central adrenal insufficiency) - peak cortisol <500nmol/L, intermediate (partial AI) - peak cortisol ≥500 nmol/L and <600 nmol/L and AS (adrenal sufficiency) - peak cortisol ≥ 600 nmol/L. In patients with diagnosed CAI HCT replacement treatment was initiated. Body weight, body fat percentage, signs, and symptoms of CAI were evaluated after 6 and 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* PWS
* age >=18 years

Exclusion Criteria:

* age <18 years
* GC treatment at last 6 months

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive patients with PWS, referred to the Department of Endocrinology Medical University of Warsaw.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
The prevalence of CAI in adult PWS patients based on HDSST. | At first visit (before HCT treatment).
  The diagnosis of CAI was based on the high-dose short Synacthen test (HDSST). The following cut-off points were used:
  1. CAI group (suspected CAI):
     • cortisol < 500 nmol/L at the 30th minute
  2. AS group (adrenal sufficiency - CAI excluded):
     • cortisol ≥ 600 nmol/L at the 30th minute
  3. Intermediate group • cortisol ≥500 nmol/L and <600 nmol/L at the 30th minute
Symptoms of CAI before hydrocortisone substitution: fatigue | Before HCT treatment
  Incidence of the fatigue in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocorisone treatment: fatigue | After 6 month HCT treatment
  Incidence of the fatigue in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocorisone treatment: fatigue | After 12 month HCT treatment
  Incidence of the fatigue in the CAI, intermediate and the AS groups.
Symptoms of CAI before hydrocortisone substitution: loss of appetite | Before HCT treatment
  Incidence of loss of appetite in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocorisone treatment: loss of appetite | After 6 month HCT treatment
  Incidence of loss of appetite in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocorisone treatment: loss of appetite | After 12 month HCT treatment
  Incidence of loss of appetite in the CAI, intermediate and the AS groups.
Symptoms of CAI before hydrocortisone substitution: muscle weakness | Before HCT treatment
  Incidence of the muscle weakness in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocortisone treatment: muscle weakness | After 6 month HCT treatment
  Incidence of the muscle weakness in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocortisone treatment: muscle weakness | After 12 month HCT treatment
  Incidence of the muscle weakness in the CAI, intermediate and the AS groups.
Symptoms of CAI before hydrocortisone substitution: myalgia | Before HCT treatment
  Incidence of the myalgia in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocorisone treatment: myalgia | After 6 month HCT treatment
  Incidence of the myalgia in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocorisone treatment: myalgia | After 12 month HCT treatment
  Incidence of the myalgia in the CAI, intermediate and the AS groups.
Symptoms of CAI before hydrocortisone substitution: arthralgia | Before HCT treatment
  Incidence of the arthralgia in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocorisone treatment: arthralgia | After 6 month HCT treatment
  Incidence of the arthralgia in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocorisone treatment: arthralgia | After 12 month HCT treatment
  Incidence of the arthralgia in the CAI, intermediate and the AS groups.
Symptoms of CAI before hydrocortisone substitution: weight loss | Before HCT treatment
  Incidence of the weight loss (>3 kg) in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocorisone treatment: weight loss | After 6 month HCT treatment
  Incidence of the weight loss (>3 kg) in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocorisone treatment: weight loss | After 12 month HCT treatment
  Incidence of the weight loss (>3 kg) in the CAI, intermediate and the AS groups.
Symptoms of CAI before hydrocortisone substitution: nausea | Before HCT treatment
  Incidence of the nausea in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocorisone treatment: nausea | After 6 month HCT treatment
  Incidence of the nausea in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocorisone treatment: nausea | After 12 month HCT treatment
  Incidence of the nausea in the CAI, intermediate and the AS groups.
Symptoms of CAI before hydrocortisone substitution: vomiting | Before HCT treatment
  Incidence of the vomiting in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocorisone treatment: vomiting | After 6 month HCT treatment
  Incidence of the vomiting in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocorisone treatment: vomiting | After 12 month HCT treatment
  Incidence of the vomiting in the CAI, intermediate and the AS groups.
Symptoms of CAI before hydrocortisone substitution: abdominal pain | Before HCT treatment
  Incidence of the abdominal pain in the CAI, intermediate and the AS groups.
Symptoms of CAI after 6 month hydrocorisone treatment: abdominal pain | After 6 month HCT treatment
  Incidence of the abdominal pain in the CAI, intermediate and the AS groups.
Symptoms of CAI after 12 month hydrocorisone treatment: abdominal pain | After 12 month HCT treatment
  Incidence of the abdominal pain in the CAI, intermediate and the AS groups.
BMI before hydrocortisone substitution in PWS patients with CAI | Before HCT treatment
  Measurement of weight and height will be combined to report BMI in kg/m^2.
BMI after 6 month hydrocortisone substitution in PWS patients with CAI | After 6 month HCT treatment
  Measurement of weight and height will be combined to report BMI in kg/m^2.
BMI after 12 month hydrocortisone substitution in PWS patients with CAI | After 12 month HCT treatment
  Measurement of weight and height will be combined to report BMI in kg/m^2.
Body fat percentage before hydrocortisone substitution in PWS patients with CAI | Before HCT treatment
  Measurement of the body fat percentage using bioelectrical impedance method.
Body fat percentage after 6 month hydrocortisone substitution in PWS patients with CAI | After 6 month HCT treatment
  Measurement of the body fat percentage using bioelectrical impedance method.
Body fat percentage after 12 month hydrocortisone substitution in PWS patients with CAI | After 12 month HCT treatment
  Measurement of the body fat percentage using bioelectrical impedance method.

SECONDARY OUTCOMES:
Concentration of morning cortisol | At first visit (before HCT treatment).
  Results of morning cortisol in the entire study group.
Concentration of ACTH | At first visit (before HCT treatment).
  Results of ACTH in the entire study group.
Concentration of dihydroepiandrosterone sulfate | At first visit (before HCT treatment).
  Results of dihydroepiandrosterone sulfate measurements in the entire study group.
Laboratory findings - short Synacthen test | At first visit (before HCT treatment).
  Results of the short Synacthen test in the entire study group.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Clinical Hospital Medical University of Warsaw, Warsaw, Poland